CLINICAL TRIAL: NCT01794611
Title: Comparison Of C-MAC Videolaryngoscopy, Kingsvision Videolaryngoscopy and Macintosh Laryngoscopy During Routine Intubation in Adult Patients
Brief Title: Different Types Of Laryngoscopes During Routine Intubation in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Guniz M.Koksal, Assoc.Prof., Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 36049
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-02

CONDITIONS: Failed or Difficult Intubation
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laryngoscopy (Experimental): Patients will be intubated by an experienced anesthesiologists. Anesthesiologist first uses Macintosh laryngoscope then KingsVision videolaryngoscope and lastly C-MAC videolaryngoscope to intubate patients. Cormack-Lehane scores, the time from the start of laryngoscopy to visualization of the vocal cords and the time from the visualization of the vocals from the successful intubation will be recorded. The success of the intubation will be assessed with bilateral chest auscultation. If visualization of the vocal cords or placing of the endotracheal tube was not successful after 60 seconds with a particular laryngoscope, it will be left out and patient will be ventilated for 1 minutes and then pass to other laryngoscopes.
  Interventions: Device: laryngoscopy

INTERVENTIONS:
Device: laryngoscopy
  Other Names: C-MAC videolaryngoscopy (Karl Storz, Tuttlingen, GERMANY); KingsVision videolaryngoscopy (KingSystems, IN, USA); Macintosh Laryngscope (Welch Allyn,USA)

SUMMARY:
C-MAC videolaryngoscope (Karl Storz, Tuttlingen, GERMANY) with its Macintosh like blade is used with standard direct laryngoscopy technique. KingsVisionTM videolaryngoscopes (KingSystems, IN, USA) have also Macintosh like single use blades that are channeled, wider and shorter than conventional Macintosh blades.We aim to compare these two laryngoscopes and Macintosh laryngoscope during routine intubation in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* 200 American Society of Anesthesiology I-III patients between 18-80 years old undergoing elective abdominal surgery and planned to be intubated orotracheally will be included in the study.

Exclusion Criteria:

* Patients with upper respiratory problems and predicted difficult airways will be excluded from the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cormack-Lehane Score | 5 minutes
  Patients will be preoxygenated with 100% oxygen for 3 minutes before the anesthesia induction. After induction when the train of four ratio reaches %0, patients will be intubated by one of three anesthesiologists with at least 10 years of experience. The anesthesiologist first will use the Macintosh laryngoscope then KingsVisionTM videolaryngoscope and lastly C-MAC videolaryngoscope to intubate the patients. The Cormack-Lehane scores observed during each laryngoscopy will be recorded

SECONDARY OUTCOMES:
time | 5 minutes
  Patients will be preoxygenated with 100% oxygen for 3 minutes before the anesthesia induction. After induction when the train of four ratio reaches %0, patients will be intubated by one of three anesthesiologists with at least 10 years of experience. The anesthesiologist first will use the Macintosh laryngoscope then KingsVisionTM videolaryngoscope and lastly C-MAC videolaryngoscope to intubate the patients. The time from the start of laryngoscopy to the visualization of the vocal cords and the time from the visualization of the vocals from the successful intubation observed during each laryngoscopy will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Guniz Koksal, Ass.Prof., Study Director — Cerrahpasa Medical Faculty Anesthesiology and Reanimation Department
Locations (1):
- Cerrahpasa Medical Faculty Anesthesiology and Reanimation Department, Istanbul, Fatih, Turkey (Türkiye)

REFERENCES:
- [Background] Xue FS, Liao X, Cheng Y. Comparative performance of C-MAC video laryngoscope and macintosh direct laryngoscope for emergency intubation. Ann Emerg Med. 2012 Dec;60(6):817-8; author reply 818-9. doi: 10.1016/j.annemergmed.2012.05.044. No abstract available. PMID 23178024